CLINICAL TRIAL: NCT03293433
Title: Quantification of microRNAs in Diagnosis of Pulmonary Nodules: Reproducibility Analysis of Intra- and Inter-observer and Inter-laboratory: Project miR-Nod
Brief Title: Quantification of microRNAs in Diagnosis of Pulmonary Nodules
Acronym: miR-Nod
Status: Completed | Type: Observational
Sponsor: University Hospital, Toulouse (Other)
Responsible Party: Sponsor
Other Study IDs: RC31/15/7818
Record Dates: First submitted 2016-07-22; First posted 2017-09-26 (Actual); Last update posted 2019-07-16 (Actual); Status verified 2019-07

CONDITIONS: Pulmonary Cancer
MeSH Terms: conditions — Lung Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Total blood punction with micro RNA exctraction
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Patient with lung cancer: Patient with pulmonary nodule showed in scanner (defined as a rounded picture higher than 5 mm and less than 30 mm in the lung parenchyma) presenting at one of the 3 participant services and meeting the inclusion criteria and exclusion. A blood punction will be performed in order to extract micro RNA.
  Interventions: Other: Blood punction

INTERVENTIONS:
Other: Blood punction — 1 blood punction during the normal pathway of care of the patient. This punction will be used to perform the extraction of micro RNA.

SUMMARY:
One of the main challenges of thoracic oncology lies in earlier diagnosis of lung cancer to improve survival rate, wich is about 15% at 5 years. This poor prognosis is often linked to late diagnosis. Efforts are being made worldwide to offer testing in patients at risk or earlier diagnosis of lung cancer in order to offer the patient curative treatments. Indeed, supported at the stage of nodule (less than 3 cm lesion), lung cancer is curable by surgery in 80% of patients. Nevertheless, there are many differential diagnoses and access to these lesions is often difficult and risky. In this context, the management of pulmonary nodules, which can be either benign lesions or beginners cancers, is a real challenge for pulmonologists and thoracic oncologists every day: it is important not to disregard a potentially operable nodule and avoiding offer patients invasive procedures for benign nodules. Indeed, many procedures (endoscopy, puncture under scanner, thoracotomy) are made to determine if suspicious nodules are benign or not. In the large National Lung Screening Trial, 28% of the procedures were associated with complications (including 11% classified severe and 16 deaths). It is therefore essential to develop non-invasive tools to refine treatment decisions.

ELIGIBILITY:
Inclusion Criteria:

* Patients with suspected abnormal chest X-ray image of malignancy defined by one solitary pulmonary nodule (NPS) NPS or 2 if operable, higher than 5 mm and less to 30 mm, without histological evidence.
* Affiliation to social security.
* Signature of informed consent.

Exclusion Criteria:

* Nodule not accessible to curative local therapy (surgery, thermoablation, radiotherapy).
* Patients in whom resection for diagnostic purposes this emergency such as one of these characters can not be delayed (these patients are not likely to belong to the people that can take a dosage of clinical interest miRNAs because the characteristics radiographic their nodule only tell them a high probability of lung cancer)
* History of an unhealed cancer
* Patients benefiting from a system of legal protection

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patient with pulmonary nodule showed in scanner (defined as a rounded picture higher than 5 mm and less than 30 mm in the lung parenchyma) presenting at one of the 3 participant services and meeting the inclusion criteria and exclusion.
Sampling Method: Non-Probability Sample
Enrollment: 103 (Actual)
Dates: Start 2015-11 (Actual); Primary Completion 2018-05 (Actual); Study Completion 2019-05 (Actual)

PRIMARY OUTCOMES:
34 micro RNA extraction as assessed by quantification of micro RNA with Real-Time Quantitative Reverse Transcription polymerase chain reaction | Through the completion of study (18 months)

SECONDARY OUTCOMES:
Measure the inter-observer reproducibility as assessed by quantification of micro RNA in total blood with Real-Time Quantitative Reverse Transcription polymerase chain reaction | Through the completion of study (18 months)
Measure the inter-laboratory reproducibility as assessed by rate of micro RNA in total blood with Real-Time Quantitative Reverse Transcription polymerase chain reaction | Through the completion of study (18 months)

CONTACTS AND LOCATIONS:
Overall Officials: GUIBERT NICOLAS, MD, Principal Investigator — University Hospital of Toulouse
Locations (2):
- France (2):
  - University Hospital of la Réunion, La Réunion
  - University Hospital of Toulouse, Toulouse

IPD SHARING:
Plan to Share IPD: Undecided